CLINICAL TRIAL: NCT00108082
Title: A Randomized, Double-Blind, Multi-Center Study Comparing the Effects of Carvedilol Modified Release Formulation (COREG MR) and Atenolol in Combination With and Compared to an Angiotensin Converting Enzyme Inhibitor (Lisinopril) on Left Ventricular Mass Regression in Hypertensive Patients With Left Ventricular Hypertrophy (LVH).
Brief Title: The CLEVER Study - Coreg And Left Ventricular Mass Regression
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: COR100216
Record Dates: First submitted 2005-04-13; First posted 2005-04-14 (Estimated); Results first posted 2009-11-09 (Estimated); Last update posted 2016-12-16 (Estimated); Status verified 2016-11

CONDITIONS: Hypertrophy, Left Ventricular
Keywords: left ventricular hypertrophy (LVH); echocardiogram; left ventricular mass regression; cardiac MRI; left ventricular mass index (LVMI)hypertension
MeSH Terms: conditions — Hypertrophy, Left Ventricular | interventions — Atenolol; Lisinopril

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Carvedilol CR (Experimental): Carvedilol controlled release (CR) 20 to 80 mg once daily (OD) plus lisinopril 20 mg OD. Participants were titrated from the starting dosage to higher dosages until their blood pressure was controlled. Participants continued to receive lisinopril 20 mg OD throughout the study. (In the protocol, carvedilol CR was referred to as carvedilol modified-release [MR].)
  Interventions: Drug: carvedilol MR; Drug: lisinopril
- Atenolol (Experimental): Atenolol 50 to 100 mg OD plus lisinopril 20 mg OD. Participants were titrated from the starting dosage to higher dosages until their blood pressure was controlled. Participants continued to receive lisinopril 20 mg OD throughout the study.
  Interventions: Drug: atenolol; Drug: lisinopril
- Lisinopril (Experimental): Lisinopril 10 to 40 mg OD plus lisinopril 20 mg OD. Participants were titrated from the starting dosage to higher dosages until their blood pressure was controlled. Participants continued to receive lisinopril 20 mg OD throughout the study.
  Interventions: Drug: lisinopril

INTERVENTIONS:
Drug: carvedilol MR — Study drug
  Other Names: Carvedilol controlled release or modified release
  Arms: Carvedilol CR
Drug: atenolol — Comparator
  Arms: Atenolol
Drug: lisinopril — Comparator
  Other Names: carvedilol MR; atenolol

SUMMARY:
This study is designed to compare the effects of COREG MR (carvedilol modified release formulation) to atenolol on indices of left ventricular dimensions when added to standardized angiotensin converting enzyme (ACE) inhibition, and to the effect of ACE inhibition alone. Subjects with LVH (left ventricular hypertrophy) and hypertension will be studied. The primary endpoint will be the change in left ventricular mass index (LVMI) characterized by magnetic resonance imaging (MRI) following 12 months of treatment. Secondary endpoints include the change in LV (left ventricular) mass, LV wall thickness, diastolic left ventricular filling parameters, and left ventricular ejection fraction by echocardiographic methods at Treatment Month 12. Composite outcomes and individual event data will also be evaluated by treatment group.

DETAILED DESCRIPTION:
A Randomized, Double-Blind, Multi-Center Study Comparing the Effects of Carvedilol Modified Release Formulation (COREG MR) and Atenolol in Combination with and Compared to an Angiotensin Converting Enzyme Inhibitor (Lisinopril) on Left Ventricular Mass Regression in Hypertensive Patients with Left Ventricular Hypertrophy (LVH).

ELIGIBILITY:
Inclusion criteria:

* Stage 1 or Stage 2 hypertension.
* Left ventricular hypertrophy.

Exclusion criteria:

* In atrial fibrillation.
* Takes beta-blocker for MI (myocardial infarction) or arrhythmia.
* Has uncontrolled diabetes, uncontrollable or symptomatic arrhythmias, unstable angina, second or third degree heart block, history of MI, COPD (chronic obstructive pulmonary disease), liver or kidney disease.
* Uses beta-2-agonists.
* Unable to undergo MRI (magnetic resonance imaging).
* Females of childbearing potential.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 287 (Actual)
Dates: Start 2005-01; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (68):
- United States (68):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Mobile, Alabama
  - GSK Investigational Site, Chandler, Arizona
  - GSK Investigational Site, Mesa, Arizona
  - GSK Investigational Site, Peoria, Arizona
  - GSK Investigational Site, Scottsdale, Arizona
  - GSK Investigational Site, Sun City, Arizona
  - GSK Investigational Site, Fresno, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Palo Alto, California
  - GSK Investigational Site, Poway, California
  - GSK Investigational Site, Sacremento, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, San Leandro, California
  - GSK Investigational Site, Santa Ana, California
  - GSK Investigational Site, Colorado Springs, Colorado
  - GSK Investigational Site, Denver, Colorado
  - GSK Investigational Site, Newark, Delaware
  - GSK Investigational Site, Washington D.C., District of Columbia
  - GSK Investigational Site, Altamonte Springs, Florida
  - GSK Investigational Site, Atlantis, Florida
  - GSK Investigational Site, Jacksonville, Florida
  - GSK Investigational Site, Kissimmee, Florida
  - GSK Investigational Site, Longwood, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Ormond Beach, Florida
  - GSK Investigational Site, Pembroke Pines, Florida
  - GSK Investigational Site, Evanston, Illinois
  - GSK Investigational Site, Vernon Hills, Illinois
  - GSK Investigational Site, Fort Wayne, Indiana
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, Scarborough, Maine
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, Columbia, Maryland
  - GSK Investigational Site, Pikesville, Maryland
  - GSK Investigational Site, Grand Rapids, Michigan
  - GSK Investigational Site, Edina, Minnesota
  - GSK Investigational Site, Minneapolis, Minnesota
  - GSK Investigational Site, Camden, New Jersey
  - GSK Investigational Site, Buffalo, New York
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Williamsville, New York
  - GSK Investigational Site, Fayetteville, North Carolina
  - GSK Investigational Site, Greensboro, North Carolina
  - GSK Investigational Site, Winston-Salem, North Carolina
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Hillsboro, Oregon
  - GSK Investigational Site, Portland, Oregon
  - GSK Investigational Site, Allentown, Pennsylvania
  - GSK Investigational Site, Camp Hill, Pennsylvania
  - GSK Investigational Site, Doylestown, Pennsylvania
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, West Grove, Pennsylvania
  - GSK Investigational Site, Warwick, Rhode Island
  - GSK Investigational Site, Columbia, South Carolina
  - GSK Investigational Site, Greenville, South Carolina
  - GSK Investigational Site, Greer, South Carolina
  - GSK Investigational Site, Kingsport, Tennessee
  - GSK Investigational Site, Knoxville, Tennessee
  - GSK Investigational Site, Nashville, Tennessee
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Danville, Virginia
  - GSK Investigational Site, Roanoke, Virginia
  - GSK Investigational Site, Springfield, Virginia
  - GSK Investigational Site, Tacoma, Washington
  - GSK Investigational Site, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Bakris GL, Tarka EA, Waterhouse B, Goulding MR, Madan A, Anderson KM, St John Sutton M, Miller AB, Reichek N. Cardiovascular risk factors in hypertension: rationale and design of studies to investigate the effects of controlled-release carvedilol on regression of left ventricular hypertrophy and lipid profile. Am J Cardiol. 2006 Oct 2;98(7A):46L-52L. doi: 10.1016/j.amjcard.2006.08.002. Epub 2006 Aug 28. PMID 17023232
- [Background] Miller AB, Reichek N, St John Sutton M, Iyengar M, Henderson LS, Tarka EA, Bakris GL. Importance of blood pressure control in left ventricular mass regression. J Am Soc Hypertens. 2010 Nov-Dec;4(6):302-10. doi: 10.1016/j.jash.2010.09.003. Epub 2010 Oct 27. PMID 20980215
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: COR100216 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: COR100216 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: COR100216 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: COR100216 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: COR100216 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: COR100216 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: COR100216 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Following screening, 413 participants were enrolled into the study to begin an open-label run-in phase with lisinopril 10 mg once daily (OD) for 1 week and then lisinopril 20 mg OD for 1 week. Of these participants, 287 were randomized to 1 of the 3 treatment regimens.
Period: Overall Study
Arm/Group | Carvedilol CR | Atenolol | Lisinopril
Started | 91 | 100 | 96
Completed | 53 (Per protocol Amendment 4, participants who had completed Month 12 prior to amendment were withdrawn.) | 68 (Per protocol Amendment 4, participants who had completed Month 12 prior to amendment were withdrawn.) | 53 (Per protocol Amendment 4, participants who had completed Month 12 prior to amendment were withdrawn.)
Not Completed | 38 | 32 | 43
Not completed — Adverse Event | 14 | 12 | 17
Not completed — Lost to Follow-up | 6 | 3 | 7
Not completed — Consent Withdrawn | 3 | 3 | 5
Not completed — Protocol Violation | 1 | 2 | 0
Not completed — Lack of Efficacy | 3 | 1 | 2
Not completed — Amendment 4: > Month 12 | 5 | 7 | 5
Not completed — Woman of Child-bearing Potential | 2 | 0 | 2
Not completed — Incorrectly Randomized | 0 | 0 | 2
Not completed — Non-compliance | 1 | 0 | 2
Not completed — Stopped Study Medication | 0 | 0 | 1
Not completed — Site Closed Study | 0 | 2 | 0
Not completed — Protocol Amendment | 0 | 1 | 0
Not completed — Study Medication Not Tapered | 0 | 1 | 0
Not completed — Subject Left Site Location | 1 | 0 | 0
Not completed — Investigator Not at Site | 1 | 0 | 0
Not completed — Blood Pressure Not Controlled | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Carvedilol CR | Atenolol | Lisinopril | Total
Number analyzed (Participants) | 91 | 100 | 96 | 287
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.6 (10.53) | 57.4 (10.95) | 55.9 (10.09) | 56.7 (10.52)
Gender [Count of Participants; unit: Participants]
  Female | 40 | 41 | 47 | 128
  Male | 51 | 59 | 49 | 159
Race/Ethnicity, Customized [Number; unit: participants]
  African American/African Heritage | 17 | 26 | 17 | 60
  American Indian/Alaska Native | 0 | 1 | 1 | 2
  Asian | 2 | 1 | 0 | 3
  White/Caucasian | 67 | 67 | 72 | 206
  Arabic/North African Heritage | 1 | 0 | 1 | 2
  Mixed Race | 1 | 0 | 1 | 2
  Not Reported | 3 | 5 | 4 | 12

OUTCOME MEASURES:

1. Primary Outcome: Model-adjusted Mean Change From Baseline in Left Ventricular Mass Indexed (LVMI) by Body Surface Area as Measured by Magnetic Resonance Imaging (MRI) at Month 12
Description: LVMI was measured by MRI at Baseline and after 12 months of treatment/Month 12. A reduction in left ventricular mass, calculated as LVMI, of 5 g/m^2 was assumed to be clinically meaningful. Change in Baseline was calculated as Month 12 value (or value after 12 months of treatment) minus the Baseline value.
Time Frame: Baseline and Month 12 (If Month 12 data were not available, the Last Observation Carried Forward [LOCF] analysis, which includes data collected on or after Month 9 of treatment to Month 12 of treatment, was used)
Population: All randomized participants who had a valid MRI at Baseline and Month 12 (LOCF on or after Month 9 to Month 12)
Measure: Mean (Standard Error); unit: grams per meters squared (g/m^2)
Arm/Group | Carvedilol CR | Atenolol | Lisinopril
Number analyzed (Participants) | 60 | 76 | 59
grams per meters squared (g/m^2) | -6.34 (0.850) | -6.67 (0.756) | -7.94 (0.850)
Statistical Analysis 1: Comparison: Carvedilol CR vs Atenolol; The null hypotheses (tested hierarchically) were that the effect of carvedilol CR + lisinopril on LV mass regression was no different than the effect of atenolol + lisinopril, and that the effect of carvedilol CR + lisinopril was no different than the effect of lisinopril + lisinopril. The primary analysis was based on an analysis of covariance (ANCOVA) with a model adjusting for treatment, stratification by hypertension class, region, and baseline value, at a 0.05 level of significance; Test type: Superiority or Other; p = 0.7651, ANCOVA; Mean Difference (Final Values) = 0.33, 95% CI [-1.83 to 2.49]
Statistical Analysis 2: Comparison: Carvedilol CR vs Lisinopril; Test type: Superiority or Other; p = 0.1711, ANCOVA; Mean Difference (Final Values) = 1.60, 95% CI [-0.70 to 3.90]

2. Secondary Outcome: Model-adjusted Mean Change From Baseline in Left Ventricular Mass Indexed by Height (LVMIH) as Measured by MRI at Month 12
Description: LVMIH was measured by MRI at Baseline and after 12 months of treatment/Month 12. Change in Baseline was calculated as Month 12 value (or value after 12 months of treatment) minus the Baseline value. LV mass depends on body size. One method of determining whether an individual has LV hypertrophy relates LV mass to height raised to a power of 2.7.
Time Frame: Baseline and Month 12 (If Month 12 data were not available, the LOCF analysis, which includes data collected on or after Month 9 of treatment to Month 12 of treatment, was used)
Population: All randomized participants who had a valid MRI at Baseline and Month 12 (LOCF on or after Month 9 to Month 12)
Measure: Mean (Standard Error); unit: g/m raised to 2.7 (g/(m^2.7))
Arm/Group | Carvedilol CR | Atenolol | Lisinopril
Number analyzed (Participants) | 60 | 76 | 59
g/m raised to 2.7 (g/(m^2.7)) | -3.19 (0.407) | -3.37 (0.361) | -3.98 (0.407)

3. Secondary Outcome: Model-adjusted Mean Change From Baseline in Left Ventricular (LV) Mass as Measured by MRI at Month 12
Description: LV Mass was measured by MRI at Baseline and after 12 months of treatment/Month 12. Change in Baseline was calculated as Month 12 value (or value after 12 months of treatment) minus the Baseline value.
Time Frame: as for outcome 2
Population: All randomized participants who had a valid MRI at Baseline and Month 12 (LOCF on or after Month 9 to Month 12)
Measure: Mean (Standard Error); unit: grams (g)
Arm/Group | Carvedilol CR | Atenolol | Lisinopril
Number analyzed (Participants) | 60 | 76 | 59
grams (g) | -13.74 (1.732) | -14.17 (1.540) | -17.17 (1.734)

4. Secondary Outcome: Model-adjusted Mean Change From Baseline in Left Ventricular Mass Indexed (LVMI) by Body Surface Area as Measured by Echocardiography at Month 12
Description: LVMI was measured by echogradiography at Baseline and after 12 months of treatment/Month 12. Change in Baseline was calculated as Month 12 value (or value after 12 months of treatment) minus the Baseline value.
Time Frame: as for outcome 2
Population: All randomized participants who had a valid echocardiogram at Baseline and Month 12 (LOCF on or after Month 9 to Month 12)
Measure: Mean (Standard Error); unit: grams per meters squared (g/m^2)
Arm/Group | Carvedilol CR | Atenolol | Lisinopril
Number analyzed (Participants) | 61 | 71 | 59
grams per meters squared (g/m^2) | -20.35 (4.027) | -20.06 (3.672) | -18.48 (3.998)

5. Secondary Outcome: Model-adjusted Mean Change From Baseline in Left Ventricular Mass Indexed by Height (LVMIH) as Measured by Echocardiography at Month 12
Description: LVMIH was measured by echogradiography at Baseline and after 12 months of treatment/Month 12. Change in Baseline was calculated as Month 12 value (or value after 12 months of treatment) minus the Baseline value.
Time Frame: Baseline and Month 12 (If Month 12 data were not available, the LOCF analysis, which includes data collected on or after Month 9 of treatment to Month 12 of treatment, was available)
Population: as for outcome 4
Measure: Mean (Standard Error); unit: g/m raised to 2.7 (g/(m^2.7))
Arm/Group | Carvedilol CR | Atenolol | Lisinopril
Number analyzed (Participants) | 61 | 71 | 59
g/m raised to 2.7 (g/(m^2.7)) | -11.78 (2.292) | -12.51 (2.100) | -11.61 (2.280)

6. Secondary Outcome: Model-adjusted Mean Change From Baseline in LV Mass as Measured by Echocardiography at Month 12
Description: LV Mass was measured by echocardiography at Baseline and after 12 months of treatment/Month 12. Change in Baseline was calculated as Month 12 value (or value after 12 months of treatment) minus the Baseline value.
Time Frame: as for outcome 2
Population: as for outcome 4
Measure: Mean (Standard Error); unit: grams
Arm/Group | Carvedilol CR | Atenolol | Lisinopril
Number analyzed (Participants) | 61 | 71 | 59
grams | -45.76 (8.338) | -40.56 (7.645) | -38.58 (8.296)

7. Secondary Outcome: Mean Change From Baseline in LV Filling Parameters as Measured by MRI at Month 12
Description: LV filling parameters, LV E-Volume and LV A-Volume, were measured by MRI at Baseline and after 12 months of treatment/Month 12. Change in Baseline was calculated as Month 12 value (or value after 12 months of treatment) minus the Baseline value. These filling parameters represent the volumes of blood filling the ventricle during the passive filling phase (E-volume) and the active filling phase caused by atrial contraction (A-volume).
Time Frame: as for outcome 2
Population: All randomized participants who had a valid MRI at Baseline and Month 12 (LOCF on or after Month 9 to Month 12)
Measure: Mean (Standard Error); unit: milliliters (mL)
Arm/Group | Carvedilol CR | Atenolol | Lisinopril
Number analyzed (Participants) | 48 | 54 | 41
milliliters (mL)
  LV E-volume | 0.364 (2.2853) | 6.763 (2.3870) | -3.406 (2.8779)
  LV A-volume | -0.513 (1.3624) | -0.565 (1.5154) | 1.088 (1.5630)

8. Secondary Outcome: Model-adjusted Mean Change From Baseline in LV End Systolic and Diastolic Volumes and Ejection Fraction as Measured by MRI at Month 12
Description: LV End Systolic and Diastolic Volumes and Ejection Fraction were measured by MRI at Baseline and after 12 months of treatment/Month 12. Change in Baseline was calculated as Month 12 value (or value after 12 months of treatment) minus the Baseline value. The ejection fraction is the fraction of the blood volume available at the end of diastole that is pumped out of the ventricules during systole.
Time Frame: as for outcome 2
Population: All randomized participants who had a valid MRI at Baseline and Month 12 (LOCF on or after Month 9 to Month 12)
Measure: Mean (Standard Error); unit: milliliters (mL)
Arm/Group | Carvedilol CR | Atenolol | Lisinopril
Number analyzed (Participants) | 60 | 76 | 59
milliliters (mL)
  LV End Systolic Volume | -1.44 (1.578) | -4.29 (1.397) | -3.04 (1.581)
  LV End Diastolic Volume | -2.86 (2.848) | -2.45 (2.522) | -7.45 (2.858)
  LV Ejection Fraction | 0.08 (0.685) | 2.16 (0.607) | -0.01 (0.685)

9. Secondary Outcome: Model-adjusted Mean Change From Baseline in LV End Systolic and Diastolic Volumes and Ejection Fraction as Measured by Echocardiography at Month 12
Description: LV End Systolic and Diastolic Volumes and Ejection Fraction were measured by echocardiography at Baseline and after 12 months of treatment/Month 12. Change in Baseline was calculated as Month 12 value (or value after 12 months of treatment) minus the Baseline value.
Time Frame: as for outcome 2
Population: as for outcome 4
Measure: Mean (Standard Error); unit: milliliters (mL)
Arm/Group | Carvedilol CR | Atenolol | Lisinopril
Number analyzed (Participants) | 60 | 76 | 59
milliliters (mL)
  LV End Systolic Volume | -3.38 (2.067) | -4.74 (1.892) | -5.34 (2.086)
  LV End Diastolic Volume | -3.07 (3.389) | -3.64 (3.108) | -9.37 (3.420)
  LV Ejection Fraction | 1.03 (0.751) | 2.33 (0.687) | 0.63 (0.756)

10. Secondary Outcome: Model-adjusted Mean Change From Baseline in Systolic and Diastolic Blood Pressure (BP) at Month 12
Description: Systolic and Diastolic BP were measured at Baseline and after 12 months of treatment/Month 12. Change in Baseline was calculated as Month 12 value (or value after 12 months of treatment) minus the Baseline value.
Time Frame: as for outcome 2
Population: All randomized participants who had a valid MRI at Baseline and Month 12 (LOCF on or after Month 9 to Month 12)
Measure: Mean (Standard Error); unit: mmHg (millimeters of mercury)
Arm/Group | Carvedilol CR | Atenolol | Lisinopril
Number analyzed (Participants) | 60 | 76 | 59
mmHg (millimeters of mercury)
  Systolic blood pressure | -21.32 (1.755) | -21.12 (1.535) | -22.53 (1.708)
  Diastolic blood pressure | -12.77 (1.103) | -14.05 (0.976) | -11.13 (1.117)

11. Secondary Outcome: Model-adjusted Ratio to Baseline as Percentage Change From Baseline in Log Transformed B-type Natriuretic Peptide (BNP) at Month 12
Description: BNP concentration (picagram per milliter) was measured at Baseline and after 12 months of treatment/Month 12. Percentage change from Baseline was based on log transformed data and was calculated as 100 x (exponent (mean change on log scale) -1) [Change is the Month 12 value (or value after 12 months of treatment) minus the Baseline value].
Time Frame: Baseline and Month 12 (If Month 12 data were not available, the LOCF was used
Population: All randomized participants who had a valid measurements at Baseline and Month 12 (LOCF)
Measure: Geometric Mean (95% Confidence Interval); unit: percentage of change
Arm/Group | Carvedilol CR | Atenolol | Lisinopril
Number analyzed (Participants) | 34 | 42 | 33
percentage of change | 51.7 [13.2 to 103.2] | 48.3 [13.0 to 94.7] | -39.1 [-54.3 to -19.0]

12. Secondary Outcome: Model-adjusted Ratio to Baseline as Percentage Change From Baseline in Log Transformed C-Reactive Protein (CRP) at Month 12
Description: CRP concentration (milligrams per deciliter) was measured at Baseline and after 12 months of treatment/Month 12. Percentage change from Baseline was based on log transformed data and calculated as 100 x (exponent (mean change on log scale) - 1). [Change in Baseline was calculated as Month 12 value (or value after 12 months of treatment) minus the Baseline value.]
Time Frame: Baseline and Month 12 (If Month 12 data were not available, the LOCF was used)
Population: All randomized participants who had a valid measurements at Baseline and Month 12 (LOCF)
Measure: Geometric Mean (95% Confidence Interval); unit: percentage of change
Arm/Group | Carvedilol CR | Atenolol | Lisinopril
Number analyzed (Participants) | 48 | 66 | 53
percentage of change | -10.63 [-27.41 to 10.02] | -3.22 [-18.82 to 15.38] | 2.70 [-15.88 to 25.37]

13. Secondary Outcome: Percentage Change From Baseline in Log Transformed Lipid Parameters at Month 12
Description: Plasma lipid concentrations (milligrams per deciliter) were measured at Baseline and after 12 months of treatment/Month 12. Percentage change from Baseline was based on log transformed data and calculated as 100 x (exponent(mean change on log scale) - 1). [Change in Baseline was calculated as Month 12 value (or value after 12 months of treatment) minus the Baseline value.]
Time Frame: Baseline and Month 12 (If Month 12 data were not available, the LOCF was used)
Population: All randomized participants who had a valid measurements at Baseline and Month 12 (LOCF)
Measure: Geometric Mean (95% Confidence Interval); unit: percentage of change
Arm/Group | Carvedilol CR | Atenolol | Lisinopril
Number analyzed (Participants) | 83 | 92 | 90
percentage of change
  Total cholesterol | 0.7 [-3.3 to 4.9] | -1.3 [-4.7 to 2.3] | -1.7 [-5.5 to 2.3]
  Low-density lipid cholesterol | 0.0 [-6.5 to 7.0] | -4.0 [-9.6 to 1.8] | -2.7 [-9.0 to 4.1]
  High-density lipid cholesterol | -4.3 [-7.7 to 0.7] | -4.7 [-7.7 to -1.6] | -1.5 [-4.9 to 2.1]
  Triglycerides | 11.0 [2.0 to 20.9] | 7.1 [-0.7 to 15.4] | 6.2 [-2.4 to 15.5]

14. Secondary Outcome: Model-adjusted Ratio to Baseline as Percentage Change From Baseline in Log Transformed Albumin Creatinine Ratio (ACR) at Month 12
Description: Urinary ACR (micrograms per milligram) was determined at Baseline and after 12 months of treatment/Month 12. Percentage change from Baseline was based on log transformed data and was calculated as 100 x (exponent (exponent (mean change on log scale) - 1. [Change in Baseline was calculated as Month 12 value (or value after 12 months of treatment) minus the Baseline value.]
Time Frame: Baseline and Month 12 (If Month 12 data were not available, the LOCF was used)
Population: All randomized participants who had a valid measurements at Baseline and Month 12 (LOCF)
Measure: Geometric Mean (95% Confidence Interval); unit: percentage of change
Arm/Group | Carvedilol CR | Atenolol | Lisinopril
Number analyzed (Participants) | 40 | 51 | 38
percentage of change | -27.1 [-39.9 to -11.6] | -20.1 [-32.4 to -5.5] | -21.5 [-35.2 to -4.8]

ADVERSE EVENTS:
Arm/Group | Carvedilol CR | Atenolol | Lisinopril
Serious Adverse Events (participants affected / at risk) | 4 | 6 | 12
Other Adverse Events (participants affected / at risk) | 54 | 61 | 52
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Carvedilol CR | Atenolol | Lisinopril
Atrial fibrillation (Cardiac disorders) | 1/91 | 0/100 | 2/96
Non-cardiac chest pain (General disorders) | 0/91 | 2/100 | 1/96
Dizziness (Nervous system disorders) | 0/91 | 0/100 | 2/96
Transient ischemic attack (Nervous system disorders) | 0/91 | 0/100 | 2/96
Abdominal pain (Gastrointestinal disorders) | 0/91 | 0/100 | 1/96
Acute coronary syndrome (Cardiac disorders) | 0/91 | 0/100 | 1/96
Chest pain (General disorders) | 0/91 | 0/100 | 1/96
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/91 | 0/100 | 1/96
Coronary artery disease (Cardiac disorders) | 1/91 | 0/100 | 0/96
Depression (Psychiatric disorders) | 1/91 | 0/100 | 0/96
Drug hypersensitivity (Immune system disorders) | 0/91 | 1/100 | 0/96
Gout (Metabolism and nutrition disorders) | 0/91 | 0/100 | 1/96
Headache (Nervous system disorders) | 0/91 | 0/100 | 1/96
Inguinal hernia obstructive (Gastrointestinal disorders) | 0/91 | 1/100 | 0/96
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0/91 | 1/100 | 0/96
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0/91 | 0/100 | 1/96
Myocardial infarction (Cardiac disorders) | 0/91 | 0/100 | 1/96
Neuropathy peripheral (Nervous system disorders) | 1/91 | 0/100 | 0/96
Pancreatitis (Gastrointestinal disorders) | 0/91 | 1/100 | 0/96
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0/91 | 0/100 | 1/96
Syncope (Nervous system disorders) | 0/91 | 0/100 | 1/96
Vision blurred (Eye disorders) | 0/91 | 0/100 | 1/96
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | Carvedilol CR | Atenolol | Lisinopril
Headache (Nervous system disorders) | 13/91 | 11/100 | 10/96
Cough (Respiratory, thoracic and mediastinal disorders) | 8/91 | 5/100 | 16/96
Dizziness (Nervous system disorders) | 13/91 | 8/100 | 6/96
Fatigue (General disorders) | 6/91 | 16/100 | 5/96
Nasopharyngitis (Infections and infestations) | 6/91 | 9/100 | 8/96
Diarrhea (Gastrointestinal disorders) | 5/91 | 7/100 | 7/96
Edema peripheral (General disorders) | 6/91 | 7/100 | 5/96
Upper respiratory tract infection (Infections and infestations) | 5/91 | 3/100 | 7/96
Muscle spasms (Musculoskeletal and connective tissue disorders) | 6/91 | 3/100 | 4/96
Bronchitis (Infections and infestations) | 6/91 | 4/100 | 2/96
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3/91 | 7/100 | 0/96

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.